CLINICAL TRIAL: NCT04935359
Title: A Randomized, Double-blind, Phase III Study, Comparing NIS793 in Combination With Gemcitabine and Nab-paclitaxel Versus (vs.) Placebo Combined With Gemcitabine and Nab-paclitaxel for First Line Treatment of Metastatic Pancreatic Ductal Adenocarcinoma (mPDAC) - daNIS-2
Brief Title: Study of Efficacy and Safety of NIS793 in Combination With Standard of Care (SOC) Chemotherapy in First-line Metastatic Pancreatic Ductal Adenocarcinoma (mPDAC) - daNIS-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNIS793B12301; 2021-000591-10 (EudraCT Number)
Record Dates: First submitted 2021-06-21; First posted 2021-06-23 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: mPDAC; NIS793; Pancreas; metastatic pancreatic ductal adenocarcinoma (mPDAC); Nab-paclitaxel; Abraxane; Gemcitabine
MeSH Terms: interventions — NIS-793; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety run-in part: NIS793+gemcitabine+nab-paclitaxel (Experimental): In the safety run-in part, participants will receive a combination of NIS793, gemcitabine and nab-paclitaxel.
  Interventions: Drug: NIS793; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Randomized part: NIS793+gemcitabine+nab-paclitaxel (Experimental): Participants will receive a combination of NIS793, gemcitabine and nab-paclitaxel
  Note: As of 07-Jul-2023, treatment with NIS793/placebo was stopped.
  Interventions: Drug: NIS793; Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Placebo
- Randomized part: placebo+gemcitabine+nab-paclitaxel (Placebo Comparator): Participants will receive a combination of placebo, gemcitabine and nab-paclitaxel
  Note: As of 07-Jul-2023, treatment with NIS793/placebo was stopped.
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Placebo

INTERVENTIONS:
Drug: NIS793 — Concentrate for solution infusion (Liquid in Vial)
  Arms: Randomized part: NIS793+gemcitabine+nab-paclitaxel; Safety run-in part: NIS793+gemcitabine+nab-paclitaxel
Drug: Nab-paclitaxel — Per locally approved formulation
Drug: Gemcitabine — Per locally approved formulation
Drug: Placebo — Dextrose 5% in water (D5W) solution for infusion
  Arms: Randomized part: NIS793+gemcitabine+nab-paclitaxel; Randomized part: placebo+gemcitabine+nab-paclitaxel

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of NIS793 in combination with gemcitabine/nab-paclitaxel versus gemcitabine/nab-paclitaxel and placebo in first-line metastatic pancreatic ductal adenocarcinoma (mPDAC).

This study aims to explore whether blockade of Transforming Growth Factor β (TGFβ) in combination with gemcitabine/nab-paclitaxel can reduce fibrosis in PDAC, restore chemo-sensitivity and ultimately lead to improvements in overall survival (OS) and other clinically relevant outcomes.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multicenter two-arm, phase III study that has two parts:

* Safety run-in part: An open-label safety run-in part will be conducted to confirm recommended phase 3 dose (RP3D) of NIS793 in combination with gemcitabine and nab-paclitaxel. Up to approximately 10 participants will be enrolled at each dose level to achieve at least 6 evaluable participants; however, if the starting dose is not recommended and a lower dose level is tested, 10 additional participants will be enrolled. The decision to open the randomized part will be based on dose confirmation and available safety, relevant PK, and other relevant data from run-in part
* Randomized part: Enrolled participants will be randomized to the two treatment arms.

The study treatment will be administered as a 28-day treatment cycle. Participants will be treated until unacceptable toxicity, disease progression per RECIST 1.1, withdrawal of consent or any other condition of treatment discontinuation specified in the protocol.

Note: As of 07-Jul-2023, treatment with NIS793/placebo was stopped. The trial was unblinded and study participants were allowed to continue with standard of care (SoC) chemotherapy (gemcitabine+ nab-paclitaxel) per investigator assessment.

ELIGIBILITY:
Inclusion Criteria:

* Applicable for both Safety run-in and Randomized part

  * Participants aged ≥18 years with histologically or cytologically confirmed (based on local assessment and per local guidelines) mPDAC eligible for treatment in the first line setting and not amenable for potentially curative surgery
  * Presence of at least one measurable lesion assessed by Computerized Tomography (CT) and/or Magnetic Resonance Imaging (MRI) according to RECIST 1.1
  * Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
  * Adequate organ function (assessed by central laboratory for eligibility)
  * Participants must have recovered from treatment-related toxicities of prior anticancer therapies to grade ≤ 1 (CTCAE v 5.0) at time of screening, except alopecia.

Main Exclusion Criteria:

* Applicable for both Safety run-in and Randomized part

  * Previous systemic anti-cancer treatment for metastatic PDAC
  * Pancreatic neuroendocrine (islet) or acinar tumors
  * Participants with known status of microsatellite instability-high (MSI-H) or mismatch repair-deficient pancreatic cancer (if status is not already available, testing is not required at screening).
  * Participant has not recovered from a major surgery performed prior to start of study treatment or has had a major surgery within 4 weeks prior to start of study treatment.
  * Radiation therapy or brain radiotherapy ≤ 4 weeks prior to start of study treatment (palliative radiotherapy to bone lesions allowed > 2 weeks prior to start of study treatment).
  * Impaired cardiac function or clinically significant cardio-vascular disease
  * Use of hematopoietic growth factors or transfusion support ≤ 2 weeks prior to start of study treatment.
  * Participant has conditions that are considered to have a high risk of clinically significant gastrointestinal tract bleeding or any other condition associated with or history of significant bleeding.
  * Serious non-healing wounds.
  * Pregnant or breast-feeding women
  * Women of childbearing potential, unless willing to use highly effective contraception methods during treatment and after stopping study treatments as indicated
  * Pre-existing peripheral neuropathy > grade 1 (CTCAE v5.0)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Safety run-in part: Percentage of participants with dose limiting toxicities (DLTs) during the first cycle (4 weeks) of treatment. | Up to 4 weeks
  Percentage of participants with DLTs during the first cycle of treatment in the safety run-in part. A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness or concomitant medication that occurs within the first cycle of treatment with NIS793 in combination with gemcitabine and nab-paclitaxel
Randomized part: Overall survival (OS) | From randomization up to death, assessed up to approximately 19 months
  OS is defined as the time from date of randomization to date of death due to any cause.

SECONDARY OUTCOMES:
Percentage of participants with Adverse Events (AEs) | Up to approximately 19 months
  Percentage of participants with AEs including changes in laboratory parameters, vital signs, body weight and cardiac assessments
Percentage of participants with dose interruptions and dose reductions of NIS793 in combination with gemcitabine and nab-paclitaxel | Up to approximately 19 months
  Tolerability measured by the percentage of participants who have dose adjustments (interruptions or reductions) of NIS793
Dose intensity of NIS793 in combination with gemcitabine and nab-paclitaxel | Up to approximately 19 months
  Tolerability measured by the dose intensity of NIS793. Dose intensity will be computed as the ratio of actual cumulative dose received and actual duration of exposure
Progression-free survival (PFS) by investigator assessment per RECIST 1.1 | From enrollment (run-in part) or randomization (randomized part) up to disease progression or death, assessed up to approximately 19 months
  PFS defined as the time from the date of enrollment (run-in part) or randomization (randomized part) to the date of the first documented progression based on investigator assessment and according to RECIST 1.1 or death due to any cause.
Overall response rate (ORR) by investigator assessment per RECIST 1.1 | Up to approximately 19 months
  ORR is defined as the proportion of participants with best overall response (BOR) of complete response (CR) or partial response (PR), as per investigator assessment and according to RECIST 1.1
Disease control rate (DCR) by investigator assessment per RECIST 1.1 | Up to approximately 19 months
  DCR is the proportion of participants with BOR of CR or PR or stable disease (SD) as per investigator assessment and according to RECIST 1.1
Time to response (TTR) by investigator assessment per RECIST 1.1 | From enrollment (run-in part) or randomization (randomized part) up to first documented response, assessed up to approximately 19 months
  TTR is defined as the duration of time between the date of enrollment (run-in part) or randomization (randomized part) and the date of first documented response of either CR or PR.
Safety run-in part: Overall Survival (OS) | From enrollment up to death, assessed up to approximately 19 months
  OS is defined as the time from the date of enrollment to date of death due to any cause.
Maximum concentration (Cmax) of NIS793 in combination with gemcitabine and nab-paclitaxel | From date of first study drug intake up to approximately 19 months
  Blood samples will be collected for analysis of Cmax of NIS793
Trough Concentration (Ctrough) of NIS793 in combination with gemcitabine and nab-paclitaxel | From date of first study drug intake up to approximately 19 months
  Blood samples will be collected for analysis of Ctrough of NIS793
Area under the curve from time zero to the last measurable concentration sampling time (AUClast) of NIS793 in combination with gemcitabine and nab-paclitaxel | From date of first study drug intake up to approximately 19 months
  Blood samples will be collected for analysis of AUClast of NIS793
Area under the curve calculated to the end of a dosing interval (tau) at steady-state (AUCtau) of NIS793 in combination with gemcitabine and nab-paclitaxel | From date of first study drug intake up to approximately 19 months
  Blood samples will be collected for analysis of AUCtau of NIS793
Time to reach maximum concentration (Tmax) of NIS793 in combination with gemcitabine and nab-paclitaxel | From date of first study drug intake up to approximately 19 months
  Blood samples will be collected for analysis of Tmax of NIS793
Randomized part: NIS793 serum concentration | From date of first study drug intake up to approximately 19 months
  Blood samples will be collected for analysis of NIS793 serum concentration
Randomized part: Anti-drug antibodies (ADA) against NIS793 prevalence at baseline | Baseline
  ADA (anti-NIS793) prevalence at baseline is defined as the proportion of participants who have an ADA positive result at baseline
Randomized part: ADA (anti-NIS793) incidence on treatment | From date of first study drug intake up to approximately 19 months
  ADA (anti-NIS793) incidence on treatment is defined as the proportion of participants who are treatment-induced ADA positive (post-baseline ADA positive with ADA-negative sample at baseline) and treatment-boosted ADA positive (post-baseline ADA positive with titer that is at least the fold titer change greater than the ADA-positive baseline titer)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (101):
- United States (9):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of California LA, Los Angeles, California
  - Advent Health Cancer Institute, Orlando, Florida
  - Fort Wayne Medical Oncology Hematology Inc, Fort Wayne, Indiana
  - NYU Clinical Cancer Center, New York, New York
  - US Oncology Research Dallas, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (2):
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Perth, Western Australia
- Belgium (4):
  - Novartis Investigative Site, Bonheiden
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Leuven
- Brazil (4):
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Ijuí, Rio Grande do Sul
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (3):
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- China (11):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Dalian, Liaoning
  - Novartis Investigative Site, Jining, Shandong
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Czechia (4):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Nový Jičín, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Prague
- Finland (2):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Tampere
- France (9):
  - Novartis Investigative Site, Nice, Alpes Maritimes
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Lyon 08
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
- Germany (7):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Halle S
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Thessaloniki, Greece
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Israel (3):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (3):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Verona, VR
- Japan (6):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Koto Ku, Tokyo
- Novartis Investigative Site, Utrecht, Netherlands
- Norway (2):
  - Novartis Investigative Site, Nordbyhagen, Oslo County
  - Novartis Investigative Site, Oslo
- Russia (2):
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Pushkin Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (3):
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Košice
- South Korea (2):
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Seoul
- Spain (4):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid
- Sweden (2):
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Umeå
- Switzerland (3):
  - Novartis Investigative Site, Bellinzona
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Sankt Gallen
- Taiwan (2):
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- United Kingdom (5):
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com